CLINICAL TRIAL: NCT03830060
Title: Clinical Usefulness of Cortisol, Antinuclear Antibodies and High-sensitivity C-reactive Protein in Diagnostic and Prognostic Evaluation of Acute Pancreatitis
Brief Title: Clinical Usefulness of Cortisol, Antinuclear Antibodies and High-sensitivity C-reactive Protein in Acute Pancreatitis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Reham I El-mahdy, Principal Investigator, Assiut University
Other Study IDs: Pancreatitis
Record Dates: First submitted 2019-02-02; First posted 2019-02-05 (Actual); Last update posted 2019-02-05 (Actual); Status verified 2019-02

CONDITIONS: Acute Pancreatitis
Keywords: Marker of inflammation; high-sensitivity CRP; Antinuclear antibodies; Cortisol
MeSH Terms: conditions — Pancreatitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group I:: Fifty AP patients on admission
  Interventions: Diagnostic Test: Measurement of cortisol
- Group II:: The previous AP patients after 72 hours
  Interventions: Diagnostic Test: Measurement of cortisol

INTERVENTIONS:
Diagnostic Test: Measurement of cortisol — Cortisol will be measured by immunofluorescence and correlated with ANA and hs-CRP

SUMMARY:
Acute pancreatitis (AP) is a potentially life-threatening disease with varying severity of presentation. Nearly 60%-80% of all cases of AP in developed countries are attributable to either gallstone disease or alcohol abuse. The incidence is similar in both sexes, although alcohol abuse is the more common cause in men and gallstones is the more common cause in women.

DETAILED DESCRIPTION:
Severe acute pancreatitis is one of the most common acute abdomens in clinical practice. Owing to its acute onset, rapid progress, and high mortality, it has become a hot clinical study spot and one of the toughest medical problems. Markers of inflammation, such as high-sensitivity CRP (hs-CRP), are predictive of the severity of acute pancreatitis and may be useful in identifying patients with severe acute pancreatitis in the early phase after onset.

Antinuclear antibodies (ANA) are important biomarkers for the autoimmune disorder. ANA may contribute to the pathogenesis of pancreatitis and ANA positivity is associated with the presence of autoimmune pancreatitis. Cortisol is released into the blood due to stimulation of corticotrophin receptors in the adrenal cortex. Thus, serum cortisol can be measured. Although the association between serum levels of some inflammatory marker and acute pancreatitis revealed, the relationship between ANA, cortisol, hs-CRP and with the severity of acute pancreatic lesions have not evaluated yet.

ELIGIBILITY:
Inclusion Criteria:

* abdominal pain consistent with AP
* serum amylase activity at least 3 times greater than the upper limit of normal
* Patients of age 18 years or more who are willing to participate in the study and give their consent for same.

Exclusion Criteria:

* Patients with severe liver disease, pulmonary embolus, sepsis, and renal failure were excluded from the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Acute pancreatitis
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-02-25 (Estimated); Primary Completion 2019-05-20 (Estimated); Study Completion 2019-05-30 (Estimated)

PRIMARY OUTCOMES:
The mean difference of cortisol before and after treatment | 72 hours
  Cortisol mean difference will be measured by immunofluorescence in acute pancreatitis.

REFERENCES:
- [Background] Zhang XP, Zhang L, Wang Y, Cheng QH, Wang JM, Cai W, Shen HP, Cai J. Study of the protective effects of dexamethasone on multiple organ injury in rats with severe acute pancreatitis. JOP. 2007 Jul 9;8(4):400-12. PMID 17625291
- [Background] Imamura T, Tanaka S, Yoshida H, Kitamura K, Ikegami A, Takahashi A, Niikawa J, Mitamura K. Significance of measurement of high-sensitivity C-reactive protein in acute pancreatitis. J Gastroenterol. 2002;37(11):935-8. doi: 10.1007/s005350200157. PMID 12483249
- [Background] Nebiker CA, Staubli S, Schafer J, Bingisser R, Christ-Crain M, Dell-Kuster S, Mueller C, Scamardi K, Viehl CT, Kolleth D, von Holzen U, Oertli D, Rosenthal R. Cortisol Outperforms Novel Cardiovascular, Inflammatory, and Neurohumoral Biomarkers in the Prediction of Outcome in Acute Pancreatitis. Pancreas. 2018 Jan;47(1):55-64. doi: 10.1097/MPA.0000000000000962. PMID 29215538
- [Background] Smyk DS, Rigopoulou EI, Koutsoumpas AL, Kriese S, Burroughs AK, Bogdanos DP. Autoantibodies in autoimmune pancreatitis. Int J Rheumatol. 2012;2012:940831. doi: 10.1155/2012/940831. Epub 2012 Jul 12. PMID 22844291